CLINICAL TRIAL: NCT02282839
Title: The Influence of Glutamine on the Side Effects of Chemo-radiation in Head and Neck Cancer Patients - A Randomized Controlled Trial
Brief Title: Oral Glutamine and Mucositis of Head and Neck Cancer Patients Undergoing Radiation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Shih-An Liu, Attending Physician, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TCVGH-1047004C
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Head and Neck Cancer; Mucositis
Keywords: Head and neck cancer; Glutamine; Oral mucositis; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Stomatitis | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Active Comparator): Oral glutamine 10 g TID (total 30 g/day) one week before radiotherapy till the end of radiotherapy
  Interventions: Dietary Supplement: Glutamine
- Control group (Placebo Comparator): Placebo (Same ingredients without glutamine) one week before radiotherapy till the end of radiotherapy
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glutamine — Powder that soluble in water for drinking, 10g TID (total 30 g per day)
  Other Names: AMINOPURE (Ajinomoto AmoniScience LLC)
  Arms: Study group
Dietary Supplement: Placebo — Powder that provided by manufacturer with the same ingredients yet without glutamine, TID use
  Arms: Control group

SUMMARY:
This study will enroll 60 consecutive patients who are scheduled to receive radiotherapy with/without chemotherapy due to head and neck cancers. Basic data will be recorded along with tumor related variables. Then they will be divided randomly into study group and control group. The study group will receive oral glutamine during radiotherapy while the control group will receive placebo during radiotherapy. The severity of oral mucositis (WHO grading system), pain status (visual analogue scale), quality of life questionnaires will also be documented. The differences between the two groups will be analyzed.

DETAILED DESCRIPTION:
Chemotherapy and radiotherapy are important therapeutic modalities for head and neck cancer patients. Oral mucositis is a common comorbidity during chemotherapy and radiotherapy. It was reported that 30-60% of patients underwent chemotherapy and over 90% of patients receiving radiotherapy had oral mucositis. Oral mucositis not only reduces the quality of life of cancer patients during therapy but also causes dysphagia and poor nutritional status. Severe oral mucositis may necessitate unplanned gaps between treatment which can undermine the chance of local control.

In terms of management of oral mucositis, maintaining of oral hygiene and avoid infection are essential manner. Topical agents such as sucralfate, benzydamine, antifungal drugs, vitamin E and treatment using laser were studied in the management of oral mucositis. Previous studies indicated the glutamine significantly reduced the incidence and severity of oral mucositis in patients underwent chemotherapy and bone marrow transplantation. However, few studies discussed the effect of glutamine on the impact of oral mucositis in head and neck cancer patients receiving radiotherapy with/without chemotherapy.

This study will enroll 60 consecutive patients who are scheduled to receive radiotherapy with/without chemotherapy due to head and neck cancers. Basic data will be recorded along with tumor related variables. Then they will be divided randomly into study group and control group. The study group will receive oral glutamine while the control group will receive placebo during radiotherapy. The severity of oral mucositis (WHO grading system, every week), pain status (visual analogue scale, every week), quality of life questionnaires (before, during and after radiotherapy) will also be documented. The differences between the two groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients scheduled to receive radiotherapy with or without chemotherapy

Exclusion Criteria:

* Prior radiotherapy to the head and neck region
* Severe liver or renal disease
* Reye's syndrome
* Allergy to glutamine
* Reluctant to join the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis | 8 weeks
  According to WHO grading system

SECONDARY OUTCOMES:
Pain status | 8 weeks
  Pain status by visual analog scale
Quality of life | 8 weeks
  Washington University Quality of life questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology Head Neck Surgery, Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Background] Bardy J, Molassiotis A, Ryder WD, Mais K, Sykes A, Yap B, Lee L, Kaczmarski E, Slevin N. A double-blind, placebo-controlled, randomised trial of active manuka honey and standard oral care for radiation-induced oral mucositis. Br J Oral Maxillofac Surg. 2012 Apr;50(3):221-6. doi: 10.1016/j.bjoms.2011.03.005. Epub 2011 Jun 1. PMID 21636188
- [Background] Wu SX, Cui TT, Zhao C, Pan JJ, Xu BY, Tian Y, Cui NJ. A prospective, randomized, multi-center trial to investigate Actovegin in prevention and treatment of acute oral mucositis caused by chemoradiotherapy for nasopharyngeal carcinoma. Radiother Oncol. 2010 Oct;97(1):113-8. doi: 10.1016/j.radonc.2010.08.003. Epub 2010 Sep 7. PMID 20826029
- [Background] Nicolatou-Galitis O, Velegraki A, Sotiropoulou-Lontou A, Dardoufas K, Kouloulias V, Kyprianou K, Kolitsi G, Skarleas C, Pissakas G, Papanicolaou VS, Kouvaris J. Effect of fluconazole antifungal prophylaxis on oral mucositis in head and neck cancer patients receiving radiotherapy. Support Care Cancer. 2006 Jan;14(1):44-51. doi: 10.1007/s00520-005-0835-2. Epub 2005 Jun 10. PMID 15947956
- [Background] Lin YS, Lin LC, Lin SW, Chang CP. Discrepancy of the effects of zinc supplementation on the prevention of radiotherapy-induced mucositis between patients with nasopharyngeal carcinoma and those with oral cancers: subgroup analysis of a double-blind, randomized study. Nutr Cancer. 2010;62(5):682-91. doi: 10.1080/01635581003605532. PMID 20574929
- [Background] Kazemian A, Kamian S, Aghili M, Hashemi FA, Haddad P. Benzydamine for prophylaxis of radiation-induced oral mucositis in head and neck cancers: a double-blind placebo-controlled randomized clinical trial. Eur J Cancer Care (Engl). 2009 Mar;18(2):174-8. doi: 10.1111/j.1365-2354.2008.00943.x. PMID 19267733
- [Background] Gautam AP, Fernandes DJ, Vidyasagar MS, Maiya AG, Nigudgi S. Effect of low-level laser therapy on patient reported measures of oral mucositis and quality of life in head and neck cancer patients receiving chemoradiotherapy--a randomized controlled trial. Support Care Cancer. 2013 May;21(5):1421-8. doi: 10.1007/s00520-012-1684-4. Epub 2012 Dec 8. PMID 23224689
- [Background] Le QT, Kim HE, Schneider CJ, Murakozy G, Skladowski K, Reinisch S, Chen Y, Hickey M, Mo M, Chen MG, Berger D, Lizambri R, Henke M. Palifermin reduces severe mucositis in definitive chemoradiotherapy of locally advanced head and neck cancer: a randomized, placebo-controlled study. J Clin Oncol. 2011 Jul 10;29(20):2808-14. doi: 10.1200/JCO.2010.32.4095. Epub 2011 Jun 13. PMID 21670453
- [Background] Ferreira PR, Fleck JF, Diehl A, Barletta D, Braga-Filho A, Barletta A, Ilha L. Protective effect of alpha-tocopherol in head and neck cancer radiation-induced mucositis: a double-blind randomized trial. Head Neck. 2004 Apr;26(4):313-21. doi: 10.1002/hed.10382. PMID 15054734
- [Background] Cerchietti LC, Navigante AH, Lutteral MA, Castro MA, Kirchuk R, Bonomi M, Cabalar ME, Roth B, Negretti G, Sheinker B, Uchima P. Double-blinded, placebo-controlled trial on intravenous L-alanyl-L-glutamine in the incidence of oral mucositis following chemoradiotherapy in patients with head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1330-7. doi: 10.1016/j.ijrobp.2006.03.042. Epub 2006 Jun 9. PMID 16765532
- [Background] Peterson DE, Jones JB, Petit RG 2nd. Randomized, placebo-controlled trial of Saforis for prevention and treatment of oral mucositis in breast cancer patients receiving anthracycline-based chemotherapy. Cancer. 2007 Jan 15;109(2):322-31. doi: 10.1002/cncr.22384. PMID 17154160
- [Background] Aquino VM, Harvey AR, Garvin JH, Godder KT, Nieder ML, Adams RH, Jackson GB, Sandler ES. A double-blind randomized placebo-controlled study of oral glutamine in the prevention of mucositis in children undergoing hematopoietic stem cell transplantation: a pediatric blood and marrow transplant consortium study. Bone Marrow Transplant. 2005 Oct;36(7):611-6. doi: 10.1038/sj.bmt.1705084. PMID 16086046